CLINICAL TRIAL: NCT02911948
Title: A Double-blinded Trial Comparing the Efficacy and Safety of Insulin Degludec/Liraglutide and Insulin Degludec Both in Combination With Metformin in Japanese Subjects With Type 2 Diabetes Mellitus Inadequately Controlled With Basal or Pre-mix/Combination Insulin Therapy and Oral Anti-diabetic Drugs
Acronym: DUAL™ II Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9068-4184; U1111-1178-3453 (Other: WHO); JapicCTI-163385 (Other: JapicCTI)
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Results first posted 2019-03-11 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec/liraglutide (Experimental)
  Interventions: Drug: Insulin degludec/liraglutide
- Insulin degludec (Active Comparator)
  Interventions: Drug: Insulin degludec

INTERVENTIONS:
Drug: Insulin degludec/liraglutide — Injected s.c. / subcutaneously (under the skin) once daily
  Arms: Insulin degludec/liraglutide
Drug: Insulin degludec — Injected s.c. / subcutaneously (under the skin) once daily
  Arms: Insulin degludec

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare the efficacy and safety of insulin degludec/liraglutide and insulin degludec both in combination with metformin in Japanese subjects with type 2 diabetes mellitus inadequately controlled with basal or pre-mix/combination insulin therapy and oral anti-diabetic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese subjects, age at least 20 years at the time of signing informed consent
* T2DM (type 2 diabetes mellitus) subjects (diagnosed clinically) for at least 6 months prior to screening
* HbA1c (glycosylated haemoglobin) 7.5-11.0 per cent [58 mmol/mol-97 mmol/mol] (both inclusive) by central laboratory analysis
* Subjects on stable daily insulin doses for at least 60 days prior to screening administered once or twice daily, either as basal insulin (e.g. IDeg, insulin glargine, insulin detemir, NPH insulin) or pre-mix/combination insulin (e.g. biphasic insulin aspart, insulin degludec/insulin aspart). Total daily insulin dose in the previous 60 days should be within 20-50 units, both inclusive, and on the day of screening, but fluctuations of plus/minus 20 per cent within the 60 days prior to screening are acceptable. The specified insulin treatment should be administered in combination with a stable daily dose of metformin within current approved Japanese label for at least 60 days prior to screening - additionally, the anti-diabetic treatment can be with or without a stable daily dose of one of the following other OADs (oral anti-diabetic drug): SU (sulfonylureas), glinides, alpha-glucosidase inhibitor, SGLT2i (sodium glucose co-transporter 2 inhibitor) or TZD (thiazolidinedione) within current approved Japanese label for at least 60 days prior to screening
* Body Mass Index (BMI) equal or above 23 kg/m^2

Exclusion Criteria:

* Receipt of any investigational medicinal product (IMP) within 30 days before screening
* Use of any anti-diabetic drug in a period of 60 days before screening (except premix/ combination or basal insulin, metformin, SU, glinides, α-GI, SGLT2i, or TZD) or anticipated change in concomitant medication, which in the investigators opinion could interfere with glucose metabolism (e.g. systemic corticosteroids or bolus insulin)
* Treatment with glucagon-like peptide-1 (GLP-1) receptor agonist during the last 60 days prior to screening and furthermore, the discontinuation of GLP-1 receptor agonist at any point in time must not have been due to safety concerns, tolerability issues or lack of efficacy, as judged by the investigator
* Treatment with dipetidyl peptidase-4 (DPP-4) inhibitors during the last 60 days prior to screening - Impaired liver function, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) equal or above 2.5 times upper limit of normal
* Renal impairment estimated Glomerular Filtration Rate (eGFR) below 60 mL/min/1.73m^2 as per Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* Screening calcitonin equal or above 50 ng/L
* History of pancreatitis (acute or chronic)
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN 2)
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (34):
- Japan (34):
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Chigasaki-shi, Kanagawa
  - Novo Nordisk Investigational Site, Chitose, Hokkaido
  - Novo Nordisk Investigational Site, Chiyoda-ku, Tokyo
  - Novo Nordisk Investigational Site, Fujisawa-shi, Kanagawa
  - Novo Nordisk Investigational Site, Fukui-shi, Fukui
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Fukuoka-shi, Fukuoka
  - Novo Nordisk Investigational Site, Fukushima
  - Novo Nordisk Investigational Site, Hokkaido
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kawagoe-shi, Saitama
  - Novo Nordisk Investigational Site, Kawaguchi-shi, Saitama
  - Novo Nordisk Investigational Site, Kumamoto
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Mitaka-shi, Tokyo
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Nagano
  - Novo Nordisk Investigational Site, Nakagami, Okinawa
  - Novo Nordisk Investigational Site, Neyagawa-shi, Osaka
  - Novo Nordisk Investigational Site, Niigata-shi, Niigata
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Saitama-shi, Saitama
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Tochigi
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Tomigusuku-shi, Okinawa
  - Novo Nordisk Investigational Site, Yamaguchi-shi, Yamaguchi

REFERENCES:
- [Result] Watada H, Kaneko S, Komatsu M, Agner BR, Nishida T, Ranthe M, Nakamura J. Superior HbA1c control with the fixed-ratio combination of insulin degludec and liraglutide (IDegLira) compared with a maximum dose of 50 units of insulin degludec in Japanese individuals with type 2 diabetes in a phase 3, double-blind, randomized trial. Diabetes Obes Metab. 2019 Dec;21(12):2694-2703. doi: 10.1111/dom.13859. Epub 2019 Sep 17. PMID 31423685
- [Result] Komatsu M, Watada H, Kaneko S, Ross Agner BF, Nishida T, Kaku K. Efficacy and safety of the fixed-ratio combination of insulin degludec and liraglutide by baseline glycated hemoglobin, body mass index and age in Japanese individuals with type 2 diabetes: A subgroup analysis of two phase III trials. J Diabetes Investig. 2021 Sep;12(9):1610-1618. doi: 10.1111/jdi.13525. Epub 2021 Mar 24. PMID 33595901
- [Derived] Watada H, Ross Agner BF, Doshi A, Bardtrum L, Ranthe MF, Billings LK. IDegLira Improves Glycemic Control in Japanese Patients with Uncontrolled Type 2 Diabetes on Premixed Insulin Therapy. Diabetes Ther. 2020 Jan;11(1):331-339. doi: 10.1007/s13300-019-00730-y. Epub 2019 Nov 23. PMID 31760599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 38 sites in Japan as follows: 38 sites screened and 37 sites randomised subjects.
Groups:
- Insulin Degludec/Liraglutide: Eligible subjects were treated with insulin degludec/liraglutide (IDegLira) in combination with metformin (at stable pre-trial dose and frequency level) for 26 weeks. The starting dose of IDegLira was 10 dose steps (10 units IDeg/0.36 mg liraglutide), with the option of choosing up to 16 dose steps (16 units IDeg/0.6 mg liraglutide) at the investigator's discretion. IDegLira was titrated twice weekly according to a predefined titration algorithm to a maximum of 50 dose steps (50 units IDeg/1.8 mg liraglutide), aiming to reach a fasting plasma glucose target between 72 mg/dL (4.0 mmol/L) and 90 mg/dL (5.0 mmol/L). IDegLira was injected subcutaneously (s.c.), once daily (OD) in the thigh, upper arm (deltoid region) or abdomen. One follow-up contact was scheduled at least 7 to 10 days after end of treatment.
- Insulin Degludec: Eligible subjects were treated with insulin degludec (IDeg) in combination with metformin (at stable pre-trial dose and frequency level) for 26 weeks. The starting dose of IDeg was 10 units IDeg, with the option of choosing up to 16 units IDeg at the investigator's discretion. IDeg was titrated twice weekly according to a predefined titration algorithm to a maximum of 50 units IDeg, aiming to reach a fasting plasma glucose target between 72 mg/dL (4.0 mmol/L) and 90 mg/dL (5.0 mmol/L). IDeg was injected subcutaneously (s.c.), once daily (OD) in the thigh, upper arm (deltoid region) or abdomen. One follow-up contact was scheduled at least 7 to 10 days after end of treatment.
Period: Overall Study
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Started | 105 | 105
Completed | 105 | 98
Not Completed | 0 | 7
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Unclassified | 0 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomised subjects (210 subjects).
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Total
Number analyzed (Participants) | 105 | 105 | 210
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (10.4) | 55.5 (10.0) | 56.0 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 42 | 77
  Male | 70 | 63 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 105 | 105 | 210
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 105 | 105 | 210
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.61 (0.88) | 8.56 (0.80) | 8.58 (0.84)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline (week 0) in HbA1c after 26 weeks of treatment.
Time Frame: week 0, week 26
Population: Full Analysis Set (FAS) included all randomised subjects (210 subjects). The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Missing data were imputed using last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Percentage of HbA1c | -1.95 (1.01) | -0.65 (0.98)
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Degludec; The response and change from baseline in response after 26 weeks are analysed using an ANCOVA model with treatment and pre-trial anti-diabetic treatment as fixed factors and corresponding baseline HbA1c value as covariate; Test type: Superiority — Superiority was considered confirmed if the upper bound of the two-sided 95% confidence interval was strictly below 0.0% for null hypothesis (H0): D=0.0% against the alternative (HA): D≠0.0%, where D is the mean difference (IDegLira - IDeg); p < 0.0001, ANCOVA; Treatment contrast = -1.28, 95% CI 2-sided [-1.50 to -1.06]

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight after 26 weeks of treatment.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Kg | -0.7 (3.5) | 0.7 (2.7)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG after 26 weeks of treatment.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
mmol/L | -2.81 (3.17) | -2.29 (2.68)

4. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose (BG) Confirmed Hypoglycaemic Episodes
Description: Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with or without symptoms consistent with hypoglycaemia.
  Severe hypoglycaemia according to the ADA definition: an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: During 26 weeks of treatment
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (210 subjects). Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: Number of episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Number of episodes | 124 | 109

5. Secondary Outcome: Daily Insulin Dose
Description: Actual daily total insulin dose after 26 weeks.
Time Frame: After 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Units | 37.6 (11.4) | 41.2 (11.5)

6. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 7.0%
Description: Number of subjects with HbA1c less than 7.0% after 26 weeks.
Time Frame: After 26 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Participants
  Yes | 75 | 23
  No | 30 | 82

7. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 7.0% and Without Weight Gain
Description: Number of subjects with HbA1c less than 7.0% and without weight gain after 26 weeks.
Time Frame: After 26 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Participants
  Yes | 50 | 9
  No | 55 | 96

8. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 7.0% Without Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment
Description: Number of subjects with HbA1c less than 7.0% after 26 weeks, who did not experience treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment.
  Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: After 26 weeks
Population: Full Analysis Set (FAS) included all randomised subjects (210 subjects). The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Missing data were imputed using last observation carried forward (LOCF) method. Number Analyzed = subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 101
Participants
  Yes | 70 | 20
  No | 35 | 81

9. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 7.0% and Without Weight Gain and Without Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment
Description: Number of subjects with HbA1c less than 7.0% and no weight gain after 26 weeks, who did not experience treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment.
  Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: After 26 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 101
Participants
  Yes | 49 | 7
  No | 56 | 94

10. Secondary Outcome: Responder (Yes/no): HbA1c Less Than or Equal to 6.5%
Description: Number of subjects with HbA1c less than or equal to 6.5% after 26 weeks.
Time Frame: After 26 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Participants
  Yes | 57 | 9
  No | 48 | 96

11. Secondary Outcome: Responder (Yes/no): HbA1c Less Than or Equal to 6.5% and Without Weight Gain
Description: Number of subjects with HbA1c less than or equal to 6.5% and without weight gain
Time Frame: After 26 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Participants
  Yes | 38 | 4
  No | 67 | 101

12. Secondary Outcome: Responder (Yes/no): HbA1c Less Than or Equal to 6.5% Without Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment
Description: Number of subjects with HbA1c less than or equal to 6.5% after 26 weeks, who did not experience treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment.
  Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: After 26 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 101
Participants
  Yes | 53 | 8
  No | 52 | 93

13. Secondary Outcome: Responder (Yes/no): HbA1c Less Than or Equal to 6.5% and Without Weight Gain and Without Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment
Description: Number of subjects with HbA1c less than or equal to 6.5% and no weight gain after 26 weeks, who did not experience treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment.
  Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: After 26 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 101
Participants
  Yes | 37 | 3
  No | 68 | 98

14. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference after 26 weeks of treatment.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
cm | -0.6 (3.8) | 0.1 (3.8)

15. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic)
Description: Change from baseline in blood pressure (systolic and diastolic) after 26 weeks of treatment.
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
mmHg
  Systolic blood pressure | -0.6 (14.7) | 0.9 (13.6)
  Diastolic blood pressure | 0.9 (9.0) | 1.2 (9.0)

16. Secondary Outcome: Self-measured Blood Glucose (SMBG) 9-point Profile (Individual Points in the Profile)
Description: Subjects were instructed to measure their plasma glucose at following timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, at bedtime, at 4:00 a.m. and before breakfast the following day.
Time Frame: After 26 weeks
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
mmol/L
  Before breakfast | 6.59 (2.32) | 6.53 (2.19)
  90 minutes after start of breakfast: number analyzed (Participants) | 103 | 103
  90 minutes after start of breakfast | 11.00 (3.67) | 12.02 (3.57)
  Before lunch: number analyzed (Participants) | 102 | 102
  Before lunch | 7.22 (2.96) | 8.49 (3.75)
  90 minutes after start of lunch: number analyzed (Participants) | 103 | 101
  90 minutes after start of lunch | 10.59 (3.17) | 12.84 (3.65)
  Before dinner: number analyzed (Participants) | 103 | 104
  Before dinner | 7.39 (2.56) | 8.60 (3.97)
  90 minutes after start of dinner: number analyzed (Participants) | 103 | 103
  90 minutes after start of dinner | 11.09 (3.24) | 13.27 (4.05)
  At Bedtime: number analyzed (Participants) | 103 | 103
  At Bedtime | 9.57 (3.54) | 11.98 (4.17)
  At 4:00 a.m.: number analyzed (Participants) | 103 | 103
  At 4:00 a.m. | 6.75 (1.98) | 7.72 (2.90)
  Before breakfast the following day: number analyzed (Participants) | 105 | 104
  Before breakfast the following day | 6.14 (1.68) | 6.40 (2.06)

17. Secondary Outcome: Change in SMBG 9-point Profile: Mean of the 9-point Profile
Description: Subjects were instructed to measure their plasma glucose at following timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, at bedtime, at 4:00 a.m. and before breakfast the following day. Mean of the 9-point profile was defined as the area under the profile (calculated using the trapezoidal method) divided by the measurement time.
Time Frame: Week 0, week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 104 | 105
mmol/L | -2.90 (2.87) | -1.11 (2.68)

18. Secondary Outcome: Change in SMBG 9-point Profile: Mean of Postprandial Plasma Glucose Increments (From Before Meal to 90 Minutes After Breakfast, Lunch and Dinner)
Description: Subjects were instructed to measure their plasma glucose at following timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, at bedtime, at 4:00 a.m. and before breakfast the following day. The mean increment over all meals was derived as the mean of all available meal increments.
Time Frame: Week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
mmol/L | -0.76 (3.00) | 0.70 (2.93)

19. Secondary Outcome: Fasting Lipid Profile
Description: Lipid profile includes total cholesterol, low density lipoprotein cholesterol (LDL cholesterol), high density lipoprotein cholesterol (HDL cholesterol), very low density lipoprotein cholesterol (VLDL cholesterol), triglycerides and free fatty acids. Lipid profile parameters are represented as ratio to baseline values.
Time Frame: Week 0, week 26
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Ratio
  Total cholesterol | 0.90 (15.9) | 0.96 (13.0)
  HDL cholesterol | 0.90 (17.5) | 0.95 (12.2)
  LDL cholesterol | 0.86 (26.7) | 0.95 (21.5)
  VLDL cholesterol | 1.02 (50.5) | 0.97 (38.2)
  Triglycerides | 1.02 (58.5) | 0.97 (39.3)
  Free fatty acids: number analyzed (Participants) | 104 | 105
  Free fatty acids | 0.86 (67.7) | 0.77 (55.3)

20. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAE)
Description: Treatment emergent adverse event is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product. If the event had onset date before the first day of exposure on randomised treatment and increased in severity during the treatment period and until 7 days after the last drug date, then this event was considered as a TEAE.
Time Frame: During 26 weeks of treatment
Population: as for outcome 4
Measure: Number; unit: Number of events
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Number of events | 280 | 210

21. Secondary Outcome: Number of Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  Severe hypoglycaemia according to the ADA definition: an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: During 26 weeks of treatment
Population: as for outcome 4
Measure: Number; unit: Number of episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Number of episodes | 52 | 43

22. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to American Diabetes Association (ADA) Definition
Description: Results represent total number of treatment emergent hypoglycaemic episodes that fall under ADA's definition of hypoglycaemia. ADA's definition of hypoglycaemia includes following categories:
  1. Severe hypoglycaemia
  2. Documented symptomatic hypoglycaemia
  3. Asymptomatic hypoglycaemia
  4. Probable symptomatic hypoglycaemia
  5. Pseudo-hypoglycaemia. Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
Time Frame: During 26 weeks of treatment
Population: as for outcome 4
Measure: Number; unit: Number of episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Number of episodes | 780 | 717

23. Secondary Outcome: Number of Treatment Emergent Nocturnal Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product. Nocturnal period: The period between 00:01 and 05:59 a.m. (both inclusive).
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  Severe hypoglycaemia according to the ADA definition: an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: During 26 weeks of treatment
Population: as for outcome 4
Measure: Number; unit: Number of episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Number of episodes | 4 | 8

24. Secondary Outcome: Change in Clinical Evaluation: Fundoscopy or Fundus Photography
Description: The result of the fundus photography/dilated fundoscopy was interpreted by the investigator into following categories: Normal; Abnormal (Abn), Not Clinically significant (NCS); Abnormal, Clinically significant (CS). Reported results are number of subjects with 'normal'; 'Abn, NCS' and 'Abn, CS' fundoscopy/fundus photography results at screening (week -2 to week 0) and week 26.
Time Frame: Screening (week -2 to week 0), week 26
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (210 subjects). Subjects in the safety set contributed to the evaluation "as treated". Missing data were imputed using last observation carried forward (LOCF) method.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Participants
  Left eye - at screening visit - normal | 53 | 70
  Left eye - at screening visit - Abn, NCS | 6 | 5
  Left eye - at screening visit - Abn, CS | 46 | 30
  Left eye - week 26 - normal | 54 | 64
  Left eye - week 26 - Abn, NCS | 7 | 7
  Left eye - week 26 - Abn, CS | 44 | 34
  Right eye - at screening visit - normal | 55 | 72
  Right eye - at screening visit - Abn, NCS | 7 | 6
  Right eye - at screening visit - Abn, CS | 43 | 27
  Right eye - week 26 - normal | 52 | 69
  Right eye - week 26 - Abn, NCS | 8 | 6
  Right eye - week 26 - Abn, CS | 45 | 30

25. Secondary Outcome: Change in Clinical Evaluation: Electrocardiogram (ECG)
Description: The result of the ECG was interpreted by the investigator into following categories: Normal; Abnormal (Abn), Not Clinically significant (NCS); Abnormal, Clinically significant (CS). Reported results are number of subjects with 'normal'; 'Abn, NCS' and 'Abn, CS' ECG results at screening (week -2 to week 0) and week 26.
Time Frame: Screening (week -2 to week 0), week 26
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Participants
  At screening visit - normal | 80 | 82
  At screening visit - Abn, NCS | 20 | 18
  At screening visit - Abn, CS | 5 | 5
  Week 26 -normal | 82 | 82
  Week 26 - Abn, NCS | 17 | 20
  Week 26 - Abn, CS | 6 | 3

26. Secondary Outcome: Change in Pulse
Description: Change in pulse after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (210 subjects). Missing data were imputed using last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
beats per minute | 6.1 (11.0) | -0.2 (7.1)

27. Secondary Outcome: Change From Baseline in Patient Reported Outcomes (PROs) of Treatment: Diabetes Therapy-Related Quality of Life (DTR-QOL)Questionnaire
Description: For the DTR-QOL questionnaire, change from baseline in the 'Total score' and the following four 'Domain scores' were analysed:
  1. Burden on social activities and daily activities
  2. Anxiety and dissatisfaction with treatment
  3. Hypoglycaemia
  4. Satisfaction with treatment. The scoring range of 'Total score' was converted to 0-100 (best case response = 100; worst case response = 0).
  The scoring range for each of four domains was converted to 0-100 (best case response = 100; worst case response = 0).
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Score on a scale
  Total score | 7.9 (14.8) | 0.1 (13.4)
  Burden on social activities and daily activities | 5.7 (17.3) | 0.6 (17.1)
  Anxiety and dissatisfaction with treatment | 12.9 (20.8) | 0.4 (17.2)
  Hypoglycaemia | -2.6 (25.5) | -1.6 (25.9)
  Satisfaction with treatment | 15.8 (22.5) | -0.4 (24.7)

28. Secondary Outcome: Change From Baseline in Patient Reported Outcomes (PROs) of Treatment: EuroQol-5D (EQ-5D-5L) Questionnaire
Description: Overall health state was rated by patients using the EQ-5D-5L visual analogue scale (VAS) and the EQ-5D-5L index score. The EQ-5D-5L VAS is a vertical scale where patients can rank their health from 0 (worst health imaginable) to 100 (best health imaginable).
  The EQ-5D-5L index score was calculated based on the 5 dimensions, i.e., mobility, self-care, usual activities (e.g., work, study), pain/discomfort and anxiety/depression with five response levels for each dimension, i.e., no problems, slight problems, moderate problems, severe problems and extreme problems. The scores from 5 dimensions are then converted to the EQ-5D-5L index score scale: 0 - 1 (full health/best-case response = 1; death/worst-case response = 0).
Time Frame: week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 105 | 105
Score on a scale
  Change in VAS score | 6.3 (17.8) | -1.0 (15.5)
  Index score | 0.02 (0.08) | -0.01 (0.11)

ADVERSE EVENTS:
Time Frame: Week 0 (randomisation) to week 26 (end of treatment) and 7 days after end of treatment.
Description: Treatment emergent adverse event is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product. If the event had onset date before the first day of exposure on randomised treatment and increased in severity during the treatment period and until 7 days after the last drug date, then this event was considered as a TEAE.
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 3/105 | 4/105
Other Adverse Events (participants affected / at risk) | 54/105 | 48/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=105) | Insulin Degludec (N=105)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=105) | Insulin Degludec (N=105)
Abdominal discomfort (Gastrointestinal disorders) | 8 (8) | 5 (5)
Constipation (Gastrointestinal disorders) | 9 (10) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 0 (0)
Diabetic retinopathy (Eye disorders) | 17 (18) | 17 (18)
Diarrhoea (Gastrointestinal disorders) | 15 (20) | 5 (6)
Nausea (Gastrointestinal disorders) | 10 (12) | 4 (5)
Viral upper respiratory tract infection (Infections and infestations) | 21 (27) | 24 (30)
Vomiting (Gastrointestinal disorders) | 9 (11) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT02911948/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT02911948/SAP_001.pdf